CLINICAL TRIAL: NCT06690489
Title: Impact of Dermatological Toxicities on Quality of Life in Patients With Early Breast Cancer Exposed to Adjuvant Endocrine Therapy: a Real-world Cross-sectional Study. BCARE (Breast Cancer Adjuvant Real-world Evaluation of Dermatological Adverse Events)
Brief Title: An Observational Real-world Study to Evaluate the Impact of Dermatological Toxicities on the Quality of Life in Patients With Early Breast Cancer Treated With Adjuvant Endocrine Therapy - BCARE (Breast Cancer Adjuvant Real-world Evaluation of Dermatological Adverse Events)
Acronym: BCARE
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS18999
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Early Breast Cancer; Skin Condition; Quality of Life
Keywords: Early breast cancer; Adjuvant endocrine therapy; Quality of life; Patient Reported Outcomes; skin toxicities
MeSH Terms: conditions — Breast Neoplasms; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this European observational study (Frane, Spain, italy, Spain and Greece) is to describe the quality of life related to dermatological toxicities, in adult women patients with Early Breast Cancer (EBC), treated with an ongoing adjuvant endocrine monotherapy initiated for 2 to 3 years ago before inclusion in the study.

In order to answer these objectives, the patient are completing 4 quality of life questionnaires focussed on dermatological issues (DLQI, Skindex-16, Hairdex and ItchyQoL) at the time of the inclusion.

Early Breast Cancer (EBC) diagnosis and history, demographics/clinical characteristics, skin care/sun protection care and skin toxicities since start of the adjuvant endocrine therapy will be collected by the investigator in the eCRF.

DETAILED DESCRIPTION:
Patients will complete the questionnaires at inclusion using a webbased PRO system

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥ 18 years at inclusion.
2. Histologically confirmed diagnosis of EBC, according to the WHO criteria and the TNM classification, at any time before inclusion.
3. Still being treated with adjuvant endocrine monotherapy, initiated 2 years (up to 1 year and 9 months) to 3 years (up to 3 years and 6 months) before the inclusion in the study.
4. Signed Informed Consent Form (ICF) or non-opposition, according to local regulations.

Exclusion Criteria:

1. Patients not able to read, understand and complete Questionnaires in local language.
2. with chronic dermatological conditions (treated or not) before initiating the adjuvant endocrine therapy that could interfere with the quality of life.
3. Patients with concomitant targeted therapies with adjuvant endocrine therapy such as CDK4/6 inhibitors or trastuzumab, and patients with ongoing treatment with neratinib.
4. Patients having relevant or severe comorbidities requiring complex therapeutic treatment.
5. Patients having a persistent post-chemotherapy alopecia (at least of grade 1)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is female patients suffering from EBC and treated with adjuvant endocrine monotherapy for 2 to 3 years, who spontaneously visit a hospital from the EADV European task force, in European countries (including France, Greece, Italy and Spain). They will be invited to participate in the study, during the inclusion period. The study population is the source population meeting eligibility criteria listed hereafter during the inclusion period.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Description of the quality-of-life data collected at the time of inclusion using the validated DLQI questionnaire | At inclusion
  The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week, including symptoms, feelings, daily activities, leisure, work, school, personal relationships, and treatment.
  The primary endpoint is the rate of patients with a DLQI score ≥ 6. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired:
  * 0 - 1 corresponds to no effect at all on patient's life,
  * 2 - 5 corresponds to small effect on patient's life,
  * 6 - 10 corresponds to moderate effect on patient's life,
  * 11 - 20 corresponds to very large effect on patient's life,
  * 21 - 30 corresponds to extremely large effect on patient's life.

SECONDARY OUTCOMES:
Quality of life data collected at the time of inclusion using the Skindex-16, Hairdex, and ItchyQoL questionnaires. | At inclusion
  The Skindex-16 includes items distributed across three domains symptoms (items 1 to 4), emotions (items 5 to 11) and functioning (items 12 to 16) and are answered on a seven-point Likert scale (varying from 0-never bothered, to 6-always bothered), which represents the frequency with which the skin problem bothered the respondent during the past week. This is a 0-100 scale, higher the score, the more quality of life is impaired.
  The Hairdex is a valuable tool for evaluating disease-specific QoL in patients with hair disorders. It consists of 48 questions across five sections: symptoms, functioning, emotions, self-confidence, and stigmatization. Each question is self-graded on a scale of 0-4, with a score of 4 indicating the most severe change from a patient's baseline quality of life.
  The ItchyQoL is a questionnaire used to measure the QoL in patients with chronic pruritus. It is composed of 22 items regarding symptoms, functions, emotions and self-perception, and is currently under
Ongoing dermatological toxicities reported by investigator according to Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0, November 2017) | At inclusion
  1. Type of toxicity
  2. Surface area involved (except for nails and oral dryness)
  3. Start date
  4. Clinical grading of the toxicity
Demographics, and clinical characteristics at the time of inclusion, including the following items | At inclusion
  1. Age, gender, weight, height
  2. Menopausal status
  3. Date of cancer diagnosis
  4. Primary tumor location
  5. T stage
  6. Prior therapies for breast cancer (type, agent name, start date, stop date)
  7. Endocrine therapy (agent name, start date) for breast cancer
  8. Current dermatological care and sun-protective behaviors

OTHER OUTCOMES:
Exploratory outcomes: History of dermatological toxicities from the beginning of current treatment to the time of inclusion | From beginning of current treatment to the time of inclusion
  1. Type of dermatological toxicity
  2. Surface area (except for nails and oral dryness)
  3. Start date and end date
  4. Grade of the toxicity, if available
  5. Change in hormonal treatment (adaptation, interruption), if applicable
Subgroups of interest | At inclusion
  * Age repartition by class (< 35 years old, 35-50, 50-65, > 65 years old)
  * Menopause status
  * Therapeutical choice before the 2/3 years of adjuvant endocrine therapy
    * Radiotherapy (yes / no)
    * Chemotherapy (yes / no), if yes, the information whether taxane was received or not will be collected
    * Adjuvant (yes/no)
    * Neoadjuvant (yes/no)
    * Target therapy (yes / no)
    * Type of adjuvant endocrine therapy
  Analyses of primary, secondary, and exploratory outcomes may be performed for some or all of these subgroups, subject to pertinence and the number of patients in each subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SIBAUD, Principal Investigator
Locations (9):
- France (2):
  - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
- Greece (2):
  - Sygros Hospital, Athens
  - Aristotle University of Thessaloniki, Thessaloniki
- Italy (3):
  - Sant'Orsola-Malpighi Hospital University of Bologna, Bologna
  - Clinica Dermatologica dell'Università di Napoli "Federico II", Napoli
  - Fondazione Policlinico A. Gemelli, Roma
- Spain (2):
  - Hospital Del Mar, Barcelona
  - Hospital General de Fuerteventura, Las Palmas

DOCUMENTS (1):
  • Study Protocol (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT06690489/Prot_000.pdf